CLINICAL TRIAL: NCT06176547
Title: Relation of Helicobacter Pylori Infection in Patients With Impaired Glucose Tolerance and Their Lipid Profile in Upper Egypt
Brief Title: Relation of Helicobacter Pylori in Prediabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled mahmmoud Ibrahim, Principal investigator, Assiut University
Other Study IDs: Relation of Helicobacter in p
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: H.Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- H.pylori in predibetic with lipid profile: Lipid profile HbA1c
  Interventions: Diagnostic Test: HbA1c

INTERVENTIONS:
Diagnostic Test: HbA1c — Blood glucose in last 3 months

SUMMARY:
The primary objective of this study is to : find the relation between H.pylori infection and pre-diabetic patients with lipid profile

. Specifically, the study aims to:

1. affect of H.pylori infection in pre-diabetic patients
2. realation between Pre-diabetic patient and lipid profile
3. Risk factor of H.pylori infection in pre-diabetic patients D)HbA1C test measures your average blood sugar level over the past 2 or 3 months.

e)Fasting Blood Sugar Test. f) the IgG antibody of h.pylori.

DETAILED DESCRIPTION:
Pre-diabetic state is aphase of impaired glucose tolerance 2 hours Postprandial Glucose (PG) in 75 g oral glucose tolerance test 140 mg/dL-199 mg/dL and/or impaired fasting glucose 100 mg/dL-125 mg/dL and/or HbA1c 5.7-6.4% [5]. Pre-diabetes is pathophysiologically similar to Type II Diabetes with basic defect being insulin resistance and early beta cell failure. The amplitude of large pulses and the rapid oscillations of insulin secretion are lost in pre-diabetes. In pre-diabetes, the glycaemic excursions are usually lower than normaland there is a delay and prolongation in the second phase of insulin secretion [6]. Recent studies have shown that colonisation with H.pylori is associated with increased development of diabetes mellitus [7-11]. A step towards identifying treatable causes of diabetes mellitus will aid the medical health system in developing new strategies in preventing the progression of pre-diabetes to overt diabetes mellitus .Dyslipidemia is a complex disease and a major risk factor foradverse cardiovascular events [12]. High levels of Low Density Lipoproteins (LDL) and low levels of High Density Lipoprotein (HDL) are associated with increased incidence of stoke and myocardial infarction [13]. dyslipidemia also plays a major role in macrovascular complications of Diabetes [14]. There is increasing evidence for the role of H.pylori infection in the initiation, development or persistence of atherosclerosis and coronary heart disease [15,16]. Therefore, exploring the role of treatable causes of dyslipidemia like H.pylorimay help in preventing the progression of dyslipidemia and its adverse effects.The present study aimed to assess the possible role of H.pylori infection on diabetic profile and lipid profile in pre-diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis ofPre-diabetic patients, age 30-60 years of either gender with fasting glucose 100 mg/dL-125 mg/dL and/or HbA1c 5.7-6.4%

Exclusion Criteria:

* insulin dependent diabetes
* hyperlipidemia

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Descriptive statistics will be used to summarize the demographic and clinical characteristics of the study population, as well as fatigue scores. Bivariate analysis (e.g., t-tests, chi-square tests) will be employed to identify significant associations between demographic, clinical, and psychosocial variables with fatigue severity.
  Multiple regression analysis will be performed to determine the independent predictors of hemodialysis-associated fatigue, considering factors with significant associations from the bivariate analysis. Statistical significance will be set at p < 0.05.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Relation of Helicobacter pylori Infection in patients with Impaired glucose tolerance and their lipid profile in upper Egypt. | Baseline
  Is there relationship between h.pylori in predibetic patients if they are positive increased to be diabetic

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Fasil, Prof, Study Director — Assiut University

REFERENCES:
- [Background] American Diabetes Association: clinical practice recommendations 1996. Diabetes Care. 1996 Jan;19 Suppl 1:S1-118. No abstract available. PMID 8689936